CLINICAL TRIAL: NCT06577350
Title: The Frequency of Osteosarcopenia and Its Relationship With Demographic and Clinical Factors in Axial Spondyloarthritis
Brief Title: Osteosarcopenia in Axial Spondyloarthritis
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ayşe A Küçükdeveci, MD, Professor, Ankara University
Other Study IDs: I11-681-21
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis; Axial Spondyloarthritis, Non-Radiographic; Osteoporosis; Sarcopenia; Osteosarcopenia
Keywords: Axial Spondyloarthritis; Ankylosing Spondylitis; Non-Radiographic Axial Spondyloarthritis; Osteoporosis; Sarcopenia; Osteosarcopenia
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis; Osteoporosis; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Axial Spondyloarthritis (AxSpA): Participants with Axial Spondyloarthritis (AxSpA)

SUMMARY:
Axial spondyloarthritis is a chronic inflammatory disease affecting the spine, sacroiliac joints, entheses, and sometimes peripheral joints with a close link to HLAB27. Typical features include inflammatory back pain, limited spinal mobility, and sacroiliitis. The term axial spondyloarthritis (AxSpA) includes both Ankylosing Spondylitis (AS) where sacroiliitis is diagnosed by X-rays, and non-radiographic AxSpA, where sacroiliitis is diagnosed via magnetic resonance imaging (MRI).

Osteoporosis is common in AS patients, and sarcopenia may also develop due to inflammation and immobilization. Osteosarcopenia, the co-occurrence of osteoporosis and sarcopenia, might have an impact on morbidity and mortality of AxSpA patients.

This cross-sectional study aims to determine the frequency of osteosarcopenia in AxSpA patients and to investigate its relationship with various demographic and clinical factors. A control group with similar age and gender distribution will be recruited to evaluate osteosarcopenia. Our hypothesis is that osteosarcopenia will be more frequent in the AxSpA group compared to the control group. The study will also identify the demographic and clinical factors associated with osteosarcopenia in AxSpa.

DETAILED DESCRIPTION:
Ankylosing Spondylitis (AS) is a chronic inflammatory disease of unknown etiology that affects the spine, sacroiliac joints, entheses regions, and sometimes peripheral joints. Its typical findings include inflammatory back pain, limited spinal mobility, and radiographic sacroiliitis. The term axial spondyloarthritis (AxSpA) describes a chronic inflammatory disease affecting the axial skeleton, including the spine and sacroiliac joints. It encompasses both patients with definite AS diagnosis with radiographic (X-ray) sacroiliitis, and patients with non-radiographic AxSpA whose sacroiliitis detected by MRI. Osteoporosis is among the clinical findings of AS. Similarly, sarcopenia may develop in AS patients due to both inflammation and immobilization. Osteosarcopenia is a clinical syndrome that includes both osteoporosis and sarcopenia. Osteosarcopenia may be a significant cause of morbidity and mortality in AxSpA patients.

This study aims to determine the frequency of osteosarcopenia in patients with AxSpA and to investigate its relationship with demographic and various clinical parameters. To determine the presence of osteoporosis, bone mineral density (BMD) measurement will be performed using Dual-energy X-ray absorptiometry (DXA). WHO definition for the diagnosis of osteoporosis will be used. A T score at or below -2.5 at the lumbal and/or hip region is defined as osteoporosis. Subsequently, to determine the presence of sarcopenia, patients will be assessed according to the European Working Group on Sarcopenia in Older People (EWGSOP2) algorithm through measurements of muscle strength, muscle mass quantity or quality, and physical performance. Skeletal muscle mass or quality will be measured by appendicular skeletal muscle mass (ASM) using both DXA, and bioelectrical impedance analysis (BIA). Skeletal muscle strength will be measured by grip strength and physical performance by gait speed. EWGSOP2 cut-off points will be used for low muscle strength (grip strength), low muscle quantity (ASM/height2) and low physical performance (gait speed). Then the sarcopenia diagnosis (probable, confirmed, severe) will be made according to the 2018 operational definition of sarcopenia by EWGSOP2. A healthy control group with similar age and gender distribution will be recruited to evaluate osteosarcopenia and compare with the patient group. After determining the presence of osteosarcopenia in AxSpA, the relationship between osteosarcopenia (sarcopenia and osteoporosis) and demographic/clinical parameters including age, gender, physical activity, disease duration, medications used (biological vs. non-biological), disease activity, spinal mobility, radiological involvement, and functional status will be investigated.

There has been no prior study on investigating osteosarcopenia in AxSpA. We expect a higher frequency osteosarcopenia in the AxSpA group compared to the control group. Additionally, the relationship between osteosarcopenia and clinical parameters will be demonstrated, thus increasing the attention and awareness of patients at high risk for developing osteosarcopenia, and facilitating early steps in treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Participants with a diagnosis of AxSpA: Participants with diagnosis of Ankylosing Spondylitis according to the modified New York criteria and participants with diagnosis of non-radiographic Spondyloarthritis (SpA) according to the Assessment of SpondyloArthritis International Society (ASAS) 2009 criteria.
* Aged 18-65 years
* Who gave consent to participate in the study

Healthy control group:

* Age- and gender-matched healthy participants (age 18-65)
* Who gave consent to participate in the study

Exclusion Criteria:

1. Systemic high-dose steroid use (>5mg/day of prednisone for more than 3 months)
2. Possible other causes of secondary sarcopenia (uncontrolled diabetes, chronic heart failure, thyroid/parathyroid disease, chronic renal failure, chronic liver failure)
3. Hand-related disorders/diseases that could affect the healthy assessment of grip strength
4. Use of any medication that could potentially affect the bone metabolism (bisphosphonates, teriparatide, anticonvulsants, heparin, and anticoagulants)
5. Psoriasis, inflammatory bowel disease
6. Infection in the thigh area where ultrasonographic evaluation will be performed
7. Body weight over 100 kg (contraindication to be positioned in the BMD device)
8. Presence of malnutrition (individuals scoring 11 or below on the Mini Nutritional Assessment-Short Form (MNA))

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include participants with AxSpA aged 18-65 years who are being followed at the Department of Physical Medicine and Rehabilitation and the Division of Rheumatology at Ankara University Faculty of Medicine.
  Age- and gender-matched healthy participants for control group will also be included. Control group will be selected from the relatives of outpatients or inpatients visiting the same clinic and from the hospital staff.
  Before the study, all participants will be asked to read the study protocol and provide written informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Presence of osteosarcopenia | 16 months
  presence of osteoporosis and sarcopenia (probable, confirmed, severe)

SECONDARY OUTCOMES:
Presence of osteoporosis | 16 months
  Presence of osteoporosis will be determined by bone mineral density (BMD) measurement using Dual-energy X-ray absorptiometry (DXA). WHO definition for the diagnosis of osteoporosis will be used. A T score at or below -2.5 at the lumbal and/or hip region is defined as osteoporosis.
Presence of sarcopenia | 16 months
  Presence of sarcopenia will be determined by EWGSOP2 algorithm through measurements of muscle strength, muscle mass quantity or quality, and physical performance. Skeletal muscle mass or quality will be measured by appendicular skeletal muscle mass (ASM) using both DXA, and bioelectrical impedance analysis (BIA). Skeletal muscle strength will be measured by grip strength and physical performance by gait speed. EWGSOP2 cut-off points will be used for low muscle strength (grip strength), low muscle quantity (ASM/height2) and low physical performance (gait speed). Then the sarcopenia diagnosis (probable, confirmed, severe) will be made according to the 2018 operational definition of sarcopenia by EWGSOP2.

OTHER OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index | 16 months
  Disease activity. Scoring 0-10, higher score indicates higher disease activity
Ankylosing Spondylitis Disease Activity Score | 16 months
  Disease activity. Scored as 4 categories: 1 inactive, 2 low disease activity, 3 high disease activity, 4 very high disease activity
Bath Ankylosing Spondylitis Metrology Index | 16 months
  Spinal mobility. Scoring 0-10, higher score indicates worse spinal mobility.
Modified Stoke Ankylosing Spondylitis Spinal Score | 16 months
  Radiological involvement. Scoring 0-72, higher score indicates more advanced radiological involvement.
Bath Ankylosing Spondylitis Functional Index | 16 months
  Functional status. Scoring 0-10, higher score indicates more physical disability.
International Physical Activity Questionnaire-short form | 16 months
  Physical activity level. Scored as 3 categories: 1 inactive, 2 minimally active, 3 active
Sonographic Thigh Adjustment Ratio | 16 months
  Regional muscle mass measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe A Küçükdeveci, MD, Principal Investigator — Ankara University, Medical Faculty
Locations (1):
- Ankara University Hospitals, Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sieper J, Braun J, Dougados M, Baeten D. Axial spondyloarthritis. Nat Rev Dis Primers. 2015 Jul 9;1:15013. doi: 10.1038/nrdp.2015.13. PMID 27188328
- [Result] Kameda H, Kobayashi S, Tamura N, Kadono Y, Tada K, Yamamura M, Tomita T. Non-radiographic axial spondyloarthritis. Mod Rheumatol. 2021 Mar;31(2):277-282. doi: 10.1080/14397595.2020.1830512. Epub 2020 Oct 12. PMID 32996809
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Result] Zhao SS, Robertson S, Reich T, Harrison NL, Moots RJ, Goodson NJ. Prevalence and impact of comorbidities in axial spondyloarthritis: systematic review and meta-analysis. Rheumatology (Oxford). 2020 Oct 1;59(Suppl4):iv47-iv57. doi: 10.1093/rheumatology/keaa246. PMID 33053193
- [Result] Magrey MN, Lewis S, Asim Khan M. Utility of DXA scanning and risk factors for osteoporosis in ankylosing spondylitis-A prospective study. Semin Arthritis Rheum. 2016 Aug;46(1):88-94. doi: 10.1016/j.semarthrit.2016.03.003. Epub 2016 Mar 9. PMID 27162010
- [Result] Klingberg E, Lorentzon M, Mellstrom D, Geijer M, Gothlin J, Hilme E, Hedberg M, Carlsten H, Forsblad-d'Elia H. Osteoporosis in ankylosing spondylitis - prevalence, risk factors and methods of assessment. Arthritis Res Ther. 2012 May 8;14(3):R108. doi: 10.1186/ar3833. PMID 22569245
- [Result] Carter S, Lories RJ. Osteoporosis: a paradox in ankylosing spondylitis. Curr Osteoporos Rep. 2011 Sep;9(3):112-5. doi: 10.1007/s11914-011-0058-z. PMID 21647573
- [Result] Barone M, Viggiani MT, Anelli MG, Fanizzi R, Lorusso O, Lopalco G, Cantarini L, Di Leo A, Lapadula G, Iannone F. Sarcopenia in Patients with Rheumatic Diseases: Prevalence and Associated Risk Factors. J Clin Med. 2018 Dec 1;7(12):504. doi: 10.3390/jcm7120504. PMID 30513782
- [Result] El Maghraoui A, Ebo'o FB, Sadni S, Majjad A, Hamza T, Mounach A. Is there a relation between pre-sarcopenia, sarcopenia, cachexia and osteoporosis in patients with ankylosing spondylitis? BMC Musculoskelet Disord. 2016 Jul 11;17:268. doi: 10.1186/s12891-016-1155-z. PMID 27401188
- [Result] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Result] Garrett S, Jenkinson T, Kennedy LG, Whitelock H, Gaisford P, Calin A. A new approach to defining disease status in ankylosing spondylitis: the Bath Ankylosing Spondylitis Disease Activity Index. J Rheumatol. 1994 Dec;21(12):2286-91. PMID 7699630
- [Result] van der Heijde D, Lie E, Kvien TK, Sieper J, Van den Bosch F, Listing J, Braun J, Landewe R; Assessment of SpondyloArthritis international Society (ASAS). ASDAS, a highly discriminatory ASAS-endorsed disease activity score in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Dec;68(12):1811-8. doi: 10.1136/ard.2008.100826. Epub 2008 Dec 5. PMID 19060001
- [Result] Yanik B, Gursel YK, Kutlay S, Ay S, Elhan AH. Adaptation of the Bath Ankylosing Spondylitis Functional Index to the Turkish population, its reliability and validity: functional assessment in AS. Clin Rheumatol. 2005 Feb;24(1):41-7. doi: 10.1007/s10067-004-0968-6. Epub 2004 Sep 8. PMID 15365877
- [Result] van der Heijde D, Landewe R, Feldtkeller E. Proposal of a linear definition of the Bath Ankylosing Spondylitis Metrology Index (BASMI) and comparison with the 2-step and 10-step definitions. Ann Rheum Dis. 2008 Apr;67(4):489-93. doi: 10.1136/ard.2007.074724. Epub 2007 Aug 29. PMID 17728332
- [Result] Creemers MC, Franssen MJ, van't Hof MA, Gribnau FW, van de Putte LB, van Riel PL. Assessment of outcome in ankylosing spondylitis: an extended radiographic scoring system. Ann Rheum Dis. 2005 Jan;64(1):127-9. doi: 10.1136/ard.2004.020503. Epub 2004 Mar 29. PMID 15051621
- [Result] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- See also: Kanis, J. A. "Assessment of osteoporosis at the primary health-care level. Technical Report." http://www. shef. ac. uk/FRAX (2008). — https://frax.shef.ac.uk/FRAX/pdfs/WHO_Technical_Report.pdf
- See also: Wenker KJ, Quint JM. Ankylosing Spondylitis. — http://www.ncbi.nlm.nih.gov/books/NBK470173/?report=reader